CLINICAL TRIAL: NCT04785144
Title: Phase 1, Open-Label, Randomized Study of the Safety and Immunogenicity of a SARS-CoV-2 Variant Vaccine (mRNA-1273.351) in Naïve and Previously Vaccinated Adults
Brief Title: Safety and Immunogenicity Study of a SARS-CoV-2 (COVID-19) Variant Vaccine (mRNA-1273.351) in Naïve and Previously Vaccinated Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-0002; 5UM1AI148373-05 (NIH)
Record Dates: First submitted 2021-03-04; First posted 2021-03-05 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2021-04-06

CONDITIONS: COVID-19; COVID-19 Immunisation
Keywords: Coronavirus; COVID-19; Immunogenicity; mRNA-1273; mRNA-1273.351; SARS-CoV-2; SARS-CoV-2 B.1.351; vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Arm 1A (Experimental): 50 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants who received two vaccinations of mRNA-1273 in DMID Protocol 20-0003 (NCT04283461). N=30.
  Interventions: Biological: mRNA-1273.351
- Arm 1B (Experimental): 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants who received two vaccinations of mRNA-1273 in DMID Protocol 20-0003 (NCT04283461). N=30.
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.351
- Arm 2A (Experimental): 100 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 57 in COVID-19 naïve participants. N=15
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.351
- Arm 2B (Experimental): 50 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 57 in COVID-19 naïve participants. N=15
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.351
- Arm 2C (Experimental): 100 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in COVID-19 naïve participants. N=20
  Interventions: Biological: mRNA-1273.351
- Arm 2D (Experimental): 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in COVID-19 naïve participants. N=20
  Interventions: Biological: mRNA-1273.351
- Arm 2E (Experimental): 100 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1, and 100 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 29 in COVID-19 naïve participants. N=20
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.351
- Arm 2F (Experimental): 50 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 29 in COVID-19 naïve participants. N=20
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.351
- Arm 2G (Experimental): 50 mcg of mRNA-1273 and 50 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in COVID-19 naïve participants. N=20
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.351
- Arm 2H (Experimental): 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in COVID-19 naïve participants. N=20
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.351

INTERVENTIONS:
Biological: mRNA-1273 — Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Arms: Arm 1B; Arm 2A; Arm 2B; Arm 2E; Arm 2F; Arm 2G; Arm 2H
Biological: mRNA-1273.351 — Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.

SUMMARY:
This is a phase 1, open-label, randomized clinical trial in males and non-pregnant females, 18 years of age and older, who are in good health, have no known history of COVID-19 or SARS-CoV-2 infection, and meet all other eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of mRNA-1273.351 manufactured by ModernaTX, Inc, given in vaccination schedules alone, sequentially, or coadministered with mRNA-1273. mRNA-1273.351 is a novel lipid nanoparticle (LNP)-encapsulated mRNA-based vaccine that encodes for a full-length, prefusion stabilized S protein of the SARS-CoV-2 B.1.351 variant. Enrollment will occur at approximately five domestic clinical research sites.

This study includes two cohorts. Cohort 1 will provide rapid information about the immunogenicity of mRNA-1273.351 in a previously vaccinated group. This cohort can inform near term public health decisions if the variant virus becomes more widespread. Cohort 2 will evaluate different strategies for generation of cross protective immune responses in a naïve population. This cohort will take longer to provide information on the immunogenicity of mRNA-1273.351, but is important to inform future public health strategies. Cohort 1 will include approximately 60 subjects 18 years of age and older who received two vaccinations of mRNA-1273 at dosages of 50 mcg, 100 mcg, or 250 mcg in the Phase 1 clinical trial (DMID 20-0003). Subjects in Cohort 1 will receive a single intramuscular (IM) injection of the designated vaccine and will be followed through 12 months after vaccination. Follow-up visits will occur on Days 8, 15, and 29, as well as 3, 6, and 12 months after the vaccination. Cohort 2 will include approximately 150 participants 18 through 55 years of age who have not received a COVID-19 vaccine, have no known history of COVID-19 or SARS-CoV-2 infection, and do not have underlying conditions that are associated with an increased risk of severe illness from SARS-CoV-2 infection. Enrollment may close before the full 150 participants based on estimates on the timing of immunogenicity results and the need to inform public health decisions. They will be randomly assigned to one of 8 treatment arms and will receive 2 or 3 IM injections of the vaccine and followed through 12 months after the last vaccination. Follow-up visits will occur 7, 14, and 28 days after each vaccination, as well as 3, 6 and 12 months post the last vaccination.

The primary objective is to evaluate the safety and reactogenicity of mRNA-1273 and mRNA-1273.351 vaccines, in naïve and previously vaccinated individuals.

DETAILED DESCRIPTION:
This is a phase 1, open-label, randomized clinical trial in males and non-pregnant females, 18 years of age and older, who are in good health, have no known history of COVID-19 or SARS-CoV-2 infection, and meet all other eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of mRNA-1273.351 manufactured by ModernaTX, Inc, given in vaccination schedules alone, sequentially, or coadministered with mRNA-1273. mRNA-1273.351 is a novel lipid nanoparticle (LNP)-encapsulated mRNA-based vaccine that encodes for a full-length, prefusion stabilized S protein of the SARS-CoV-2 B.1.351 variant. Enrollment will occur at approximately five domestic clinical research sites.

This study includes two cohorts. Cohort 1 will provide rapid information about the immunogenicity of mRNA-1273.351 in a previously vaccinated group. This cohort can inform near term public health decisions if the variant virus becomes more widespread. Cohort 2 will evaluate different strategies for generation of cross protective immune responses in a naïve population. This cohort will take longer to provide information on the immunogenicity of mRNA-1273.351, but is important to inform future public health strategies. Cohort 1 will include approximately 60 subjects 18 years of age and older who received two vaccinations of mRNA-1273 at dosages of 50 mcg, 100 mcg, or 250 mcg in the Phase 1 clinical trial (DMID 20-0003). Subjects in Cohort 1 will receive a single intramuscular (IM) injection of the designated vaccine and will be followed through 12 months after vaccination. Follow-up visits will occur on Days 8, 15, and 29, as well as 3, 6, and 12 months after the vaccination. Cohort 2 will include approximately 150 participants 18 through 55 years of age who have not received a COVID-19 vaccine, have no known history of COVID-19 or SARS-CoV-2 infection, and do not have underlying conditions that are associated with an increased risk of severe illness from SARS-CoV-2 infection. Enrollment may close before the full 150 participants based on estimates on the timing of immunogenicity results and the need to inform public health decisions. They will be randomly assigned to one of 8 treatment arms and will receive 2 or 3 IM injections of the vaccine and followed through 12 months after the last vaccination. Follow-up visits will occur 7, 14, and 28 days after each vaccination, as well as 3, 6 and 12 months post the last vaccination.

The primary objective is to evaluate the safety and reactogenicity of mRNA-1273 and mRNA-1273.351 vaccines, in naïve and previously vaccinated individuals. The secondary objective is to assess humoral immunogenicity of mRNA-1273 and mRNA-1273.351 vaccines, in naïve and previously vaccinated individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent prior to initiation of any study procedures.
2. Be able to understand and agrees to comply with planned study procedures and be available for all study visits.
3. Agrees to the collection of venous blood per protocol.
4. Cohort 1: previously received 2 doses of mRNA-1273 intramuscular (IM) as part of DMID 20-0003.
5. Cohort 1: Male or non-pregnant female, >/= 18 years of age at time of enrollment. Cohort 2: Male or non-pregnant female, 18 through 55 years of age at time of enrollment.
6. Women of childbearing potential* must agree to practice abstinence or use at least one acceptable primary form of contraception.**, *** Note: These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).

   * Not of childbearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure(R) placement).

   ** Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the subject's first vaccination, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products.

   *** Must use at least one acceptable primary form of contraception for at least 30 days prior to the first vaccination and at least one acceptable primary form of contraception for 60 days after the last vaccination.
7. In good health.*

   * As determined by medical history and physical examination to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of subjects. Chronic medical diagnoses/conditions should be stable for the last 60 days (no hospitalizations, emergency room, or urgent care for condition or need for supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 60 days before enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome or for dose optimization, as determined by the participating site PI or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity, and do not indicate a worsening of medical diagnosis/condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided the change was not precipitated by deterioration in the chronic medical condition, and there is no anticipated additional risk to the subject or interference with the evaluation of responses to study vaccination.
8. Oral temperature is less than 100.0 degrees Fahrenheit (37.8 degrees Celsius).
9. Must agree to have samples stored for secondary research.
10. Agrees to adhere to Lifestyle Considerations throughout study duration.
11. Must agree to refrain from donating blood or plasma during the study (outside of this study).

Exclusion Criteria:

1. Positive pregnancy test prior to each vaccine administration.
2. BMI > 40.0 kg / m^2.
3. Female subject who is breastfeeding.
4. Has any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes study participation.*

   * Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
5. Presence of self-reported or medically documented significant medical or psychiatric condition(s).*

   * Significant medical or psychiatric conditions include but are not limited to: Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma) requiring daily medications currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years. Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics.

   Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), history of myocarditis or pericarditis as an adult, myocardial infarction (MI) within past 6 months, coronary artery bypass surgery or stent placement, or uncontrolled cardiac arrhythmia.

   Neurological or neurodevelopmental conditions (e.g., history of migraines in the past 5 years, epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease).

   Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.

   An autoimmune disease, including hypothyroidism without a defined non-autoimmune cause, localized or history of psoriasis.

   An immunodeficiency of any cause. Chronic kidney disease, estimated glomerular filtration rate (eGFR) < 60 mL / min / 1.73m^2.

   Type 2 diabetes mellitus, not including prediabetes.
6. Has an acute illness*, as determined by the participating site PI or appropriate sub-investigator, with or without fever [oral temperature >/= 38.0 degrees Celsius (100.4 degrees Fahrenheit)] within 72 hours prior to each vaccination.

   * An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
7. Has participated in another investigational study involving any investigational product* within 5 half-lives before the first vaccine administration.

   * study drug, biologic or device.
8. Currently enrolled in or plans to participate in another clinical trial with an investigational agent* that will be received during the study-reporting period.**

   * Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.

   ** Up to 15 months after the first vaccination.
9. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to drugs or any previous licensed or unlicensed vaccines or to polyethylene glycol (PEG) or a PEG-containing product.
10. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness.*

    * Including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs during the preceding 6-month period prior to vaccine administration (Day 1). The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.
11. Anticipating the need for immunosuppressive treatment within the next 6 months.
12. Received immunoglobulins and/or any blood or blood products within the 4 months before the first vaccine administration or at any time during the study.
13. Has any blood dyscrasias or significant disorder of coagulation.
14. Received or plans to receive a licensed, live vaccine within 4 weeks before or after each vaccination.
15. Received or plans to receive a licensed, inactivated vaccine within 2 weeks before or after each vaccination.
16. Receipt of any other SARS-CoV-2 vaccine or any experimental coronavirus vaccine at any time prior to or during the study, except Cohort 1 subjects who received mRNA-1273 in DMID 20-0003.
17. Close contact of anyone known to have SARS-CoV-2 infection within 14 days prior to vaccine administration.
18. History of COVID-19 diagnosis, positive SARS-CoV-2 PCR test, or, for Cohort 2 only, a known positive SARS-CoV-2 serologic test.
19. On current treatment with investigational agents for prophylaxis of COVID-19.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The Hope Clinic of Emory University, Decatur, Georgia
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington

REFERENCES:
- [Derived] Anderson E, Jackson L, Rouphael N, Widge A, Montefiori D, Doria-Rose N, Suthar M, Cohen K, O'Connell S, Makowski M, Makhene M, Buchanan W, Spearman P, Creech CB, O'Dell S, Schmidt S, Leav B, Bennett H, Pajon R, Posavad C, Hural J, Beigel J, Albert J, Abebe K, Eaton A, Rostad C, Rebolledo P, Kamidani S, Graciaa D, Coler R, McDermott A, Ledgerwood J, Mascola J, DeRosa S, Neuzil K, McElrath MJ, Roberts P. Safety and Immunogenicity of a Third Dose of SARS-CoV-2 mRNA Vaccine - An Interim Analysis. Res Sq [Preprint]. 2022 May 3:rs.3.rs-1222037. doi: 10.21203/rs.3.rs-1222037/v1. PMID 35547849

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited for this study include males and non-pregnant females of 18 or more years of age, who were in good health, had no known history of COVID-19 or SARS-CoV-2 infection, and met all other eligibility criteria. Participants were recruited from the Phase 1 clinical trial (NCT04283461) and from the community surrounding the clinical sites. Enrollment occurred between 31MAR2021 and 27MAY2021.
Groups:
- Arm 1A: 50 mcg of mRNA-1273.351: 50 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants who received two vaccinations of mRNA-1273.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Participants were recruited from a Phase 1 clinical trial (NCT04283461).
- Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351: 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants who received two vaccinations of mRNA-1273.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Participants were recruited from a Phase 1 clinical trial (NCT04283461).
- Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351: 100 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 57.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Participants were recruited from the community surrounding the clinical sites.
- Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351: 50 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 57.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Participants were recruited from the community surrounding the clinical sites.
- Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351: 100 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Participants were recruited from the community surrounding the clinical sites.
- Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351: 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Participants were recruited from the community surrounding the clinical sites.
- Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351: 100 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1, and 100 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 29.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
- Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351: 50 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 29.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Participants were recruited from the community surrounding the clinical sites.
- Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351: 50 mcg of mRNA-1273 and 50 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Participants were recruited from the community surrounding the clinical sites.
- Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351: 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  mRNA-1273.351: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the pre fusion stabilized spike protein of the B.1.351 variant SARS-CoV-2 strain. mRNA-1273.351 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.
  Participants were recruited from the community surrounding the clinical sites.
Period: Overall Study
Arm/Group | Arm 1A: 50 mcg of mRNA-1273.351 | Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Started | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13
Completed | 20 | 22 | 5 | 6 | 11 | 9 | 9 | 10 | 8 | 10
Not Completed | 5 | 1 | 0 | 0 | 1 | 4 | 4 | 2 | 5 | 3
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 4 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Unable to continue due to work schedule | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1A: 50 mcg of mRNA-1273.351: 50 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants who received two vaccinations of mRNA-1273.
- Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351: 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants who received two vaccinations of mRNA-1273.
- Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351: 100 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 57.
- Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351: 50 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 57.
- Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351: 100 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
- Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351: 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
- Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351: 100 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1, and 100 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 29.
- Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351: 50 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 29.
- Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351: 50 mcg of mRNA-1273 and 50 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
- Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351: 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
- Total: Total of all reporting groups
Arm/Group | Arm 1A: 50 mcg of mRNA-1273.351 | Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | Total
Number analyzed (Participants) | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (19.0) | 43.7 (17.0) | 39.2 (14.0) | 40.3 (11.9) | 39.1 (11.5) | 35.8 (13.0) | 32.7 (9.8) | 36.1 (10.8) | 34.9 (11.4) | 36.7 (10.0) | 39.2 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 3 | 3 | 3 | 5 | 6 | 8 | 6 | 6 | 63
  Male | 14 | 11 | 2 | 3 | 9 | 8 | 7 | 4 | 7 | 7 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 9
  Not Hispanic or Latino | 21 | 22 | 5 | 6 | 11 | 12 | 11 | 12 | 12 | 13 | 125
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 1 | 2 | 2 | 2 | 2 | 1 | 3 | 3 | 2 | 19
  White | 21 | 22 | 2 | 4 | 7 | 11 | 9 | 9 | 10 | 10 | 105
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13 | 135
Height [Mean (Standard Deviation); unit: centimeters] | 171.62 (7.60) | 172.70 (11.39) | 170.44 (8.96) | 175.10 (10.27) | 177.44 (10.13) | 175.30 (13.25) | 173.22 (11.16) | 169.83 (10.44) | 178.17 (9.88) | 175.08 (8.14) | 173.75 (10.17)
Weight [Mean (Standard Deviation); unit: kilograms] | 73.68 (13.68) | 76.40 (13.10) | 78.44 (19.60) | 72.13 (12.53) | 81.43 (17.92) | 83.19 (21.04) | 74.53 (21.89) | 84.59 (21.19) | 87.53 (17.54) | 88.42 (19.65) | 79.66 (17.82)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.86 (3.27) | 25.53 (3.12) | 27.30 (8.13) | 23.47 (2.97) | 25.77 (4.73) | 26.76 (4.56) | 24.34 (4.80) | 29.09 (5.78) | 27.47 (4.54) | 28.85 (6.28) | 26.23 (4.74)
Time Between Previous Trial Dose and Dose 1 [Mean (Standard Deviation); unit: Days] — Population: Participants in Arms 1A-B were recruited from a previous trial (NCT04283461) and were administered a booster dose in this trial. Thus, they had varying times between the previous trial dose and dose 1 administration. Arms 2A-H were naïve participants and had a set schedule between doses.
  Days
    number analyzed (Participants) | 25 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 48
    (all) | 321.4 (24.8) | 319.4 (25.7) |  |  |  |  |  |  |  |  | 320.5 (25.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Medically-attended Adverse Events (MAAEs)
Description: Number of participants that experienced MAAEs during the course of the study.
Time Frame: Day 1 to study completion, up to 1 year post last dose
Population: The Safety Analysis Population includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: 50 mcg of mRNA-1273.351 | Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13
Participants | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Frequency of Any New-onset Chronic Medical Conditions (NOCMCs)
Description: Number of participants that experienced any NOCMCs during the course of the study.
Time Frame: Day 1 to study completion, up to 1 year post last dose
Population: The Safety Analysis Population includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: 50 mcg of mRNA-1273.351 | Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13
Participants | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Frequency of Any Protocol Specified Adverse Events of Special Interest (AESIs)
Description: Number of participants that experienced any AESIs during the course of the study. An adverse event of special interest (serious or non-serious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor is required. AESIs include anosmia, ageusia, subacute thyroiditis, acute pancreatitis, appendicitis, rhabdomyolysis, acute respiratory distress syndrome, coagulation disorders, acute cardiovascular injury, acute kidney injury, acute liver injury, dermatologic findings, multisystem inflammatory disorders, thrombocytopenia, acute aseptic arthritis, new onset of or worsening of neurologic disease, anaphylaxis, and other syndromes.
Time Frame: Day 1 to study completion, up to 1 year post last dose
Population: The Safety Analysis Population includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: 50 mcg of mRNA-1273.351 | Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13
Participants | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Frequency of Any Serious Adverse Events (SAEs)
Description: The number of participants that experience any SAEs from Day 1 to study completion. An AE or suspected adverse reaction is considered serious if, in the view of either the participating site PI or appropriate sub-investigator or the sponsor, it results in: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 to study completion, up to 1 year post last dose
Population: The Safety Analysis Population includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351: 50 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 29.
- 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351: 50 mcg of mRNA-1273 and 50 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
- 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351: 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
Arm/Group | Arm 1A: 50 mcg of mRNA-1273.351 | Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Frequency of Solicited Reactogenicity Adverse Events (AEs)
Description: The number of participants that experienced at least one solicited (local and systemic) AE through 7 days post vaccination. Systemic events include: fatigue, headache, myalgia, arthralgia, nausea, chills and fever. Local events include: pain at injection site, erythema, and induration.
Time Frame: Day 1 through Day 7 for Arms 1A-2H, Day 29 through Day 36 for Arms 2A-2H, Day 57-64 for Arms 2A-2B
Population: The Safety Analysis Population includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- 1A: 50 mcg of mRNA-1273.351: 50 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants who received two vaccinations of mRNA-1273.
- 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351: 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants who received two vaccinations of mRNA-1273.
- 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351: 100 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 57.
- 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351: 50 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29, and 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 57.
- 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351: 100 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
- 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351: 50 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
- 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351: 100 mcg mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1, and 100 mcg mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid on Day 29.
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13
Participants
  Local Events | 24 | 20 | 5 | 6 | 10 | 12 | 13 | 11 | 12 | 13
  Systemic Events | 22 | 20 | 5 | 6 | 12 | 11 | 12 | 11 | 12 | 12

6. Primary Outcome: Grade of Solicited Reactogenicity Adverse Events (AEs)
Description: Number of participants who experienced any solicited (local and systemic) AEs through 7 days post vaccination by grade. Systemic events include: fatigue, headache, myalgia, arthralgia, nausea, chills and fever. Local events include: pain at injection site, erythema, and induration.
Time Frame: Day 1 through Day 7 for Arms 1A-2H, Day 29 through Day 36 for Arms 2A-2H, Day 57-64 for Arms 2A-2B
Population: The Safety Analysis Population includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13
Participants
  None | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Mild | 4 | 6 | 0 | 2 | 2 | 3 | 1 | 2 | 1 | 4
  Moderate | 18 | 13 | 2 | 4 | 6 | 7 | 8 | 7 | 9 | 6
  Severe | 2 | 3 | 3 | 0 | 4 | 2 | 4 | 2 | 3 | 3

7. Primary Outcome: Frequency of Unsolicited Adverse Events (AEs) by Relationship to Study Product
Description: Number of events of any unsolicited AE through 28 days post vaccination by relationship to study product and severity, experienced by participants in the Safety Analysis population. Unsolicited AEs were events that were spontaneously reported by the subject, or revealed by observation, physical examination or other diagnostic procedures.
Time Frame: Day 1 through Day 29 for Arms 1A-2H, Day 29 through Day 57 for Arms 2A-2H, Day 57 through Day 85 from Arms 2A-2B
Population: The Safety Analysis population includes all participants who received one dose of vaccine.
Measure: Number; unit: Events
Groups:
- 2F: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351: 25 mcg of mRNA-1273 and 25 mcg of mRNA-1273.351 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29.
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | 2F: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13
Events
  Not Related | 10 | 11 | 4 | 5 | 6 | 0 | 3 | 6 | 7 | 8
  Related | 12 | 3 | 3 | 1 | 5 | 16 | 4 | 2 | 13 | 10

8. Primary Outcome: Grade of Any Unsolicited Adverse Events (AEs)
Description: Number of any unsolicited AEs through 28 days post vaccination by severity.
Time Frame: Day 1 through Day 29 for Arms 1A-2H, Day 29 through Day 57 for Arms 2A-2H, Day 57 through Day 85 from Arms 2A-2B
Population: The Safety Analysis Population includes all participants who received one dose of vaccine.
Measure: Number; unit: Events
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23 | 5 | 6 | 12 | 13 | 13 | 12 | 13 | 13
Events
  Mild | 14 | 7 | 4 | 4 | 9 | 11 | 4 | 4 | 15 | 5
  Moderate | 6 | 6 | 3 | 2 | 1 | 5 | 3 | 3 | 5 | 10
  Severe | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3

9. Secondary Outcome: Geometric Mean Titer (GMT) of Antibody Against WA-1 S2-P for Arms 1A and 1B
Description: Geometric mean titer (GMT) of antibody against WA-1 S2-P using a 4-plex ECLIA Assay.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 366
Population: The modified intent-to-treat (mITT) population includes all participants who received one dose of vaccine and contributed both pre- and at least one post-vaccination venous blood samples for immunogenicity testing for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23
Titer
  Day 1, Pre-Booster Dose | 40555.5 [29458.3 to 55833.2] | 35988.3 [28423.6 to 45566.3]
  Day 15 | 1065642.8 [831651.5 to 1365469.3] | 993561.1 [808666.6 to 1220730.1]
  Day 29 | 1276347.8 [996652.8 to 1634534.8] | 1169728.7 [935192.8 to 1463083.6]
  Day 91 | 660179.8 [482539.5 to 903216.0] | 623572.3 [476570.8 to 815917.4]
  Day 181: number analyzed (Participants) | 22 | 23
  Day 181 | 335476.6 [225669.7 to 498713.5] | 320314.1 [236469.5 to 433887.4]
  Day 366: number analyzed (Participants) | 20 | 22
  Day 366 | 287835.1 [175517.5 to 472027.2] | 268030.8 [165874.5 to 433101.5]

10. Secondary Outcome: Geometric Mean Titer (GMT) of Antibody Against WA-1 S2-P for Arms 2A and 2B
Description: Geometric mean titer (GMT) of antibody against WA-1 S2-P using a 4-plex ECLIA Assay.
Time Frame: Day 1 Pre-Dose, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 147, Day 237, Day 422
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351
Number analyzed (Participants) | 5 | 6
Titer
  Day 1, Pre-Dose | 1687.1 [7.1 to 399625.2] | 601.5 [35.0 to 10335.2]
  Day 15 | 408309.5 [42298.5 to 3941435.8] | 103325.5 [15879.5 to 672322.4]
  Day 29 | 348738.5 [58387.7 to 2082947.7] | 85622.2 [15912.6 to 460715.8]
  Day 43 | 1028488.1 [427257.0 to 2475764.6] | 622864.8 [369077.3 to 1051163.4]
  Day 57 | 689051.1 [311987.0 to 1521830.7] | 440293.4 [252560.9 to 767570.3]
  Day 71 | 687273.1 [354218.2 to 1333484.0] | 485649.5 [319892.3 to 737296.4]
  Day 85 | 565917.9 [329154.7 to 972986.3] | 373198.2 [263014.4 to 529540.9]
  Day 147 | 254433.8 [141392.1 to 457851.2] | 144121.2 [102293.2 to 203052.9]
  Day 237 | 66652.9 [32372.9 to 137232.1] | 37379.9 [26884.8 to 51972.0]
  Day 422: number analyzed (Participants) | 5 | 5
  Day 422 | 86226.1 [13571.1 to 547849.5] | 254786.0 [67095.1 to 967520.6]

11. Secondary Outcome: Geometric Mean Titer (GMT) of Antibody Against WA-1 S2-P for Arms 2C-H
Description: Geometric mean titer (GMT) of antibody against WA-1 S2-P using a 4-plex ECLIA Assay
Time Frame: Day 1 Pre-Dose, Day 15, Day 29, Day 43, Day 57, Day 119, Day 209, Day 394
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 12 | 13 | 13 | 12 | 13 | 12
Titer
  Day 1, Pre-Dose | 271.4 [56.6 to 1301.5] | 92.3 [44.2 to 193.1] | 346.7 [106.4 to 1129.4] | 645.6 [131.8 to 3162.9] | 159.8 [66.1 to 386.6] | 192.7 [85.3 to 435.2]
  Day 15 | 30368.1 [12103.4 to 76194.9] | 21710.7 [8990.4 to 52429.1] | 156640.9 [49419.1 to 496495.6] | 91564.4 [23858.3 to 351410.3] | 67811.1 [33999.0 to 135249.3] | 62111.1 [21508.0 to 179365.2]
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 11 | 12 | 12
  Day 29 | 28662.2 [12663.2 to 64874.5] | 25301.5 [11770.7 to 54386.3] | 125557.3 [43644.1 to 361209.1] | 118461.4 [42867.4 to 327360.8] | 63247.3 [30848.1 to 129674.8] | 73048.1 [31225.8 to 170885.1]
  Day 43: number analyzed (Participants) | 11 | 12 | 12 | 11 | 12 | 12
  Day 43 | 225186.6 [179455.3 to 282571.7] | 258723.7 [177985.0 to 376087.6] | 550894.5 [307970.4 to 985435.0] | 427940.0 [296902.0 to 616811.9] | 433732.7 [321427.9 to 585275.9] | 313325.4 [142344.2 to 689686.0]
  Day 57: number analyzed (Participants) | 12 | 12 | 12 | 10 | 12 | 12
  Day 57 | 171256.0 [129663.6 to 226190.2] | 184762.6 [131348.8 to 259897.5] | 380485.7 [199113.7 to 727069.0] | 320340.2 [213401.9 to 480866.6] | 301884.2 [214565.4 to 424738.1] | 321259.8 [233943.1 to 441166.4]
  Day 119: number analyzed (Participants) | 12 | 12 | 11 | 10 | 9 | 12
  Day 119 | 78575.3 [57452.9 to 107463.4] | 86821.0 [62315.8 to 120962.7] | 176619.9 [91660.5 to 340327.6] | 142765.3 [79953.4 to 254922.7] | 142664.0 [86638.7 to 234918.3] | 134238.4 [99246.4 to 181567.8]
  Day 209: number analyzed (Participants) | 11 | 12 | 12 | 9 | 9 | 11
  Day 209 | 33582.4 [20553.9 to 54869.3] | 32839.3 [24068.6 to 44806.1] | 71377.9 [38729.6 to 131548.1] | 43724.8 [26058.5 to 73367.7] | 44229.8 [22017.3 to 88851.7] | 40884.3 [26065.6 to 64127.4]
  Day 394: number analyzed (Participants) | 11 | 9 | 8 | 10 | 8 | 9
  Day 394 | 234021.1 [118055.7 to 463898.6] | 77061.1 [19964.5 to 297449.5] | 399456.3 [136582.2 to 1168273.1] | 218022.7 [129671.7 to 366571.2] | 347444.1 [124288.7 to 971266.2] | 499494.9 [217234.3 to 1148507.2]

12. Secondary Outcome: Geometric Mean Titer (GMT) of Antibody Against B.1.351 S2-P for Arms 1A and 1B
Description: Geometric Mean Titer (GMT) of Antibody Against B.1.351 S2-P using a 4-plex ECLIA Assay.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 366
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23
Titer
  Day 1, Pre-Booster Dose | 16714.5 [12487.0 to 22373.1] | 14513.9 [11417.0 to 18451.0]
  Day 15 | 598971.7 [463182.5 to 774569.7] | 465312.9 [377354.5 to 573773.7]
  Day 29 | 633384.7 [495342.5 to 809896.5] | 495722.6 [399293.1 to 615439.9]
  Day 91 | 334468.3 [248187.1 to 450744.8] | 279134.2 [214470.3 to 363294.7]
  Day 181: number analyzed (Participants) | 22 | 23
  Day 181 | 158501.6 [109437.9 to 229561.9] | 136205.1 [100841.4 to 183970.2]
  Day 366: number analyzed (Participants) | 20 | 22
  Day 366 | 131964.9 [82509.5 to 211063.5] | 119198.6 [73758.3 to 192633.4]

13. Secondary Outcome: Geometric Mean Titer (GMT) of Antibody Against B.1.351 S2-P for Arms 2A and 2B
Description: Geometric Mean Titer (GMT) of Antibody Against B.1.351 S2-P using a 4-plex ECLIA Assay.
Time Frame: Day 1 Pre-Dose, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 147, Day 237, Day 422
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351
Number analyzed (Participants) | 5 | 6
Titer
  Day 1, Pre-Dose | 733.5 [2.4 to 225877.7] | 328.9 [22.3 to 4844.4]
  Day 15 | 244620.3 [19555.8 to 3059912.2] | 54497.0 [8122.1 to 365658.8]
  Day 29 | 192969.1 [27809.7 to 1338997.0] | 39611.5 [6922.0 to 226679.9]
  Day 43 | 402295.2 [143809.2 to 1125389.9] | 195404.8 [103020.2 to 370636.7]
  Day 57 | 277548.7 [108735.7 to 708445.2] | 142696.8 [72199.7 to 282028.5]
  Day 71 | 310800.9 [148772.2 to 649295.8] | 192337.7 [117452.4 to 314968.3]
  Day 85 | 264416.1 [141960.4 to 492502.6] | 152131.5 [102734.3 to 225280.1]
  Day 147 | 115520.5 [54985.1 to 242702.0] | 56873.6 [41022.8 to 78849.1]
  Day 237 | 37901.7 [14721.7 to 97579.8] | 17270.3 [13122.3 to 22729.4]
  Day 422 | 46726.0 [8400.5 to 259904.3] | 113969.3 [32167.4 to 403794.5]

14. Secondary Outcome: Geometric Mean Titer (GMT) of Antibody Against B.1.351 S2-P for Arms 2C-H
Description: Geometric Mean Titer (GMT) of Antibody Against B.1.351 S2-P using a 4-plex ECLIA Assay.
Time Frame: Day 1 Pre-Dose, Day 15, Day 29, Day 43, Day 57, Day 119, Day 209, Day 394
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 12 | 13 | 13 | 12 | 13 | 12
Titer
  Day 1, Pre-Dose | 197.8 [46.2 to 846.0] | 47.3 [15.8 to 141.8] | 229.3 [71.9 to 731.7] | 267.5 [51.9 to 1377.8] | 63.8 [20.3 to 200.6] | 104.4 [39.9 to 273.3]
  Day 15 | 26421.7 [10770.1 to 64818.6] | 19904.5 [7952.6 to 49819.2] | 96043.2 [34594.5 to 266641.0] | 37894.4 [9601.4 to 149559.6] | 44484.5 [21394.3 to 92495.4] | 44725.5 [15959.5 to 125340.2]
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 11 | 12 | 12
  Day 29 | 26830.7 [12625.6 to 57018.0] | 23453.5 [10893.1 to 50496.9] | 70695.1 [27514.5 to 181641.9] | 45830.5 [15820.3 to 132768.7] | 42977.0 [20315.3 to 90917.8] | 50232.1 [21540.3 to 117141.6]
  Day 43: number analyzed (Participants) | 11 | 12 | 12 | 11 | 12 | 12
  Day 43 | 307328.7 [254174.5 to 371598.7] | 344899.3 [246574.6 to 482432.3] | 291453.2 [162217.6 to 523648.3] | 212624.2 [139205.5 to 324764.6] | 357231.6 [267417.1 to 477211.1] | 255274.4 [113042.9 to 576462.3]
  Day 57: number analyzed (Participants) | 12 | 12 | 12 | 10 | 12 | 12
  Day 57 | 224236.3 [186925.2 to 268994.9] | 251732.7 [188930.7 to 335410.6] | 209943.5 [113481.0 to 388402.1] | 161775.1 [100793.2 to 259652.2] | 252862.2 [186024.0 to 343715.4] | 257459.9 [193904.8 to 341846.2]
  Day 119: number analyzed (Participants) | 12 | 12 | 11 | 10 | 9 | 12
  Day 119 | 107644.5 [85403.5 to 135677.5] | 127871.2 [95537.2 to 171148.3] | 105382.0 [55465.4 to 200221.5] | 80663.9 [44544.0 to 146072.8] | 115540.1 [74664.1 to 178794.3] | 104319.3 [76850.4 to 141606.4]
  Day 209: number analyzed (Participants) | 11 | 12 | 12 | 9 | 9 | 11
  Day 209 | 53366.1 [35371.4 to 80515.3] | 51958.2 [38148.2 to 70767.3] | 47486.8 [27079.6 to 83272.9] | 28167.4 [17107.2 to 46378.1] | 39447.9 [21334.5 to 72940.0] | 32817.3 [21453.7 to 50200.0]
  Day 394: number analyzed (Participants) | 11 | 9 | 8 | 10 | 8 | 9
  Day 394 | 208767.5 [104731.8 to 416147.6] | 83893.8 [26424.9 to 266345.4] | 259147.4 [92939.4 to 722593.2] | 135964.4 [76772.8 to 240792.7] | 266166.9 [98556.9 to 718821.7] | 331123.7 [148034.1 to 740659.9]

15. Secondary Outcome: Number of Participants Who Seroconverted Against WA-1 S2-P for Arms 1A and 1B
Description: Number of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against WA-1 S2-P.
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 366
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23
Participants
  Day 15 | 25 | 23
  Day 29 | 25 | 23
  Day 91 | 24 | 22
  Day 181: number analyzed (Participants) | 22 | 23
  Day 181 | 19 | 18
  Day 366: number analyzed (Participants) | 20 | 22
  Day 366 | 16 | 13

16. Secondary Outcome: Number of Participants Who Seroconverted Against WA-1 S2-P for Arms 2A and 2B
Description: Number of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against WA-1 S2-P.
Time Frame: Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 147, Day 237, Day 422
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351
Number analyzed (Participants) | 5 | 6
Participants
  Day 15 | 4 | 6
  Day 29 | 4 | 6
  Day 43 | 4 | 6
  Day 57 | 4 | 6
  Day 71 | 4 | 6
  Day 85 | 4 | 6
  Day 147 | 4 | 6
  Day 237 | 3 | 5
  Day 422: number analyzed (Participants) | 5 | 5
  Day 422 | 3 | 5

17. Secondary Outcome: Number of Participants Who Seroconverted Against WA-1 S2-P for Arms 2C-H
Description: Number of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against WA-1 S2-P.
Time Frame: Day 15, Day 29, Day 43, Day 57, Day 119, Day 209, Day 394
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 12 | 13 | 13 | 12 | 13 | 12
Participants
  Day 15 | 11 | 13 | 13 | 12 | 13 | 12
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 11 | 12 | 12
  Day 29 | 11 | 13 | 13 | 11 | 12 | 12
  Day 43: number analyzed (Participants) | 11 | 12 | 12 | 11 | 12 | 12
  Day 43 | 11 | 12 | 12 | 11 | 12 | 12
  Day 57: number analyzed (Participants) | 12 | 12 | 12 | 10 | 12 | 12
  Day 57 | 11 | 12 | 12 | 10 | 12 | 12
  Day 119: number analyzed (Participants) | 12 | 12 | 11 | 10 | 9 | 12
  Day 119 | 11 | 12 | 11 | 10 | 9 | 12
  Day 209: number analyzed (Participants) | 11 | 12 | 12 | 9 | 9 | 11
  Day 209 | 11 | 12 | 12 | 9 | 9 | 11
  Day 394: number analyzed (Participants) | 11 | 9 | 8 | 10 | 8 | 9
  Day 394 | 11 | 9 | 8 | 10 | 8 | 9

18. Secondary Outcome: Number of Participants Who Seroconverted Against B.1.351 S2-P for Arms 1A and 1B
Description: Number of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against B.1.351 S2-P.
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 366
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23
Participants
  Day 15 | 25 | 23
  Day 29 | 25 | 23
  Day 91 | 25 | 23
  Day 181: number analyzed (Participants) | 22 | 23
  Day 181 | 20 | 18
  Day 366: number analyzed (Participants) | 20 | 22
  Day 366 | 18 | 15

19. Secondary Outcome: Number of Participants Who Seroconverted Against B.1.351 S2-P for Arms 2A and 2B
Description: as for outcome 18
Time Frame: Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 147, Day 237, Day 422
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351
Number analyzed (Participants) | 5 | 6
Participants
  Day 15 | 4 | 6
  Day 29 | 4 | 6
  Day 43 | 4 | 6
  Day 57 | 4 | 6
  Day 71 | 4 | 6
  Day 85 | 4 | 6
  Day 147 | 4 | 5
  Day 237 | 3 | 5
  Day 422: number analyzed (Participants) | 5 | 5
  Day 422 | 3 | 5

20. Secondary Outcome: Number of Participants Who Seroconverted Against B.1.351 S2-P for Arms 2C-H
Description: as for outcome 18
Time Frame: Day 15, Day 29, Day 43, Day 57, Day 119, Day 209, Day 394
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 12 | 13 | 13 | 12 | 13 | 12
Participants
  Day 15 | 11 | 13 | 13 | 12 | 13 | 12
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 11 | 12 | 12
  Day 29 | 11 | 13 | 13 | 11 | 12 | 12
  Day 43: number analyzed (Participants) | 11 | 12 | 12 | 11 | 12 | 12
  Day 43 | 11 | 12 | 12 | 11 | 12 | 12
  Day 57: number analyzed (Participants) | 12 | 12 | 12 | 10 | 12 | 12
  Day 57 | 11 | 12 | 12 | 10 | 12 | 12
  Day 119: number analyzed (Participants) | 12 | 12 | 11 | 10 | 9 | 12
  Day 119 | 11 | 12 | 11 | 10 | 9 | 12
  Day 209: number analyzed (Participants) | 11 | 12 | 12 | 9 | 9 | 11
  Day 209 | 11 | 12 | 12 | 9 | 9 | 11
  Day 394: number analyzed (Participants) | 11 | 9 | 8 | 10 | 8 | 9
  Day 394 | 11 | 9 | 8 | 10 | 8 | 9

21. Secondary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G for Arms 1A and 1B
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 366
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23
Titer
  Day 1, Pre-Booster Dose | 127.0 [96.1 to 167.8] | 114.9 [87.9 to 150.3]
  Day 15 | 2111.4 [1615.0 to 2760.3] | 2460.4 [1952.2 to 3100.8]
  Day 29 | 2544.6 [1872.3 to 3458.3] | 2829.8 [2112.4 to 3790.9]
  Day 91 | 3175.5 [2124.4 to 4746.6] | 3572.8 [2668.0 to 4784.5]
  Day 181: number analyzed (Participants) | 22 | 23
  Day 181 | 1623.6 [1045.0 to 2522.6] | 1794.5 [1198.6 to 2686.6]
  Day 366: number analyzed (Participants) | 20 | 22
  Day 366 | 749.6 [422.1 to 1331.1] | 653.8 [308.4 to 1386.2]

22. Secondary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G for Arms 2A and 2B
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G
Time Frame: Day 1 Pre-Dose, Day 29, Day 57, Day 85, Day 147, Day 237, Day 422
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351
Number analyzed (Participants) | 5 | 6
Titer
  Day 1, Pre-Dose | 37.2 [4.3 to 318.7] | 9.4 [4.0 to 21.7]
  Day 29 | 1587.5 [72.4 to 34798.3] | 135.5 [15.9 to 1156.8]
  Day 57 | 3759.4 [1566.5 to 9022.1] | 2600.2 [1296.4 to 5215.2]
  Day 85 | 3046.9 [1732.8 to 5357.7] | 1875.4 [776.3 to 4530.8]
  Day 147 | 1855.5 [931.1 to 3697.7] | 705.8 [377.1 to 1320.8]
  Day 237 | 484.8 [200.0 to 1175.2] | 120.9 [62.8 to 232.8]
  Day 422: number analyzed (Participants) | 5 | 5
  Day 422 | 604.0 [77.6 to 4700.2] | 1372.1 [313.1 to 6012.4]

23. Secondary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G for Arms 2C-H
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against D614G. Arms 2C and 2G Day 43 samples were used for pseudovirus neutralization assay validation and results included for completeness. Samples for other vaccination groups at Day 43 were not tested for neutralization.
Time Frame: Day 1 Pre-Dose, Day 29, Day 43, Day 57, Day 119, Day 209, Day 394
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 12 | 13 | 13 | 12 | 13 | 12
Titer
  Day 1, Pre-Dose | 10.8 [3.2 to 36.5] | 5.3 [4.6 to 6.2] | 12.5 [5.9 to 26.6] | 12.1 [5.3 to 27.5] | 6.8 [4.6 to 9.9] | 12.7 [3.5 to 46.4]
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 11 | 12 | 12
  Day 29 | 24.1 [6.5 to 89.8] | 16.0 [5.3 to 48.0] | 357.3 [93.1 to 1372.0] | 366.9 [88.2 to 1525.8] | 89.9 [29.0 to 278.5] | 102.7 [21.2 to 497.4]
  Day 43: number analyzed (Participants) | 10 | 0 | 0 | 0 | 12 | 0
  Day 43 | 316.9 [161.2 to 622.9] |  |  |  | 1926.4 [1099.7 to 3374.6] |
  Day 57: number analyzed (Participants) | 12 | 12 | 12 | 10 | 12 | 12
  Day 57 | 280.8 [141.1 to 558.6] | 313.6 [162.7 to 604.4] | 1914.4 [895.5 to 4092.3] | 939.9 [395.9 to 2231.7] | 1316.6 [725.9 to 2388.1] | 2017.1 [939.4 to 4331.1]
  Day 119: number analyzed (Participants) | 12 | 12 | 11 | 10 | 9 | 12
  Day 119 | 178.6 [86.1 to 370.7] | 147.6 [82.3 to 264.5] | 1042.3 [486.4 to 2233.8] | 476.1 [182.6 to 1241.3] | 749.9 [326.4 to 1722.8] | 938.9 [393.3 to 2241.4]
  Day 209: number analyzed (Participants) | 11 | 12 | 12 | 9 | 9 | 11
  Day 209 | 113.1 [56.0 to 228.6] | 85.2 [51.6 to 140.8] | 497.5 [222.9 to 1110.1] | 183.2 [63.7 to 527.4] | 272.2 [98.9 to 749.0] | 315.0 [114.8 to 863.8]
  Day 394: number analyzed (Participants) | 11 | 9 | 8 | 10 | 8 | 9
  Day 394 | 863.1 [354.7 to 2100.3] | 179.8 [33.8 to 957.8] | 1793.5 [670.6 to 4796.8] | 1091.6 [605.4 to 1968.1] | 2265.8 [480.4 to 10686.0] | 2958.7 [1677.1 to 5219.7]

24. Secondary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351 for Arms 1A and 1B
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351.
Time Frame: Day 1 Pre-Booster Dose, Day 15, Day 29, Day 91, Day 181, Day 366
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23
Titer
  Day 1, Pre-Booster Dose | 23.2 [16.4 to 32.6] | 24.2 [17.3 to 33.7]
  Day 15 | 1100.1 [867.3 to 1395.5] | 864.6 [665.9 to 1122.5]
  Day 29 | 1773.8 [1306.2 to 2408.8] | 1326.1 [916.0 to 1919.7]
  Day 91 | 1150.2 [761.5 to 1737.5] | 792.8 [537.9 to 1168.5]
  Day 181: number analyzed (Participants) | 22 | 23
  Day 181 | 482.0 [295.0 to 787.5] | 367.7 [220.7 to 612.8]
  Day 366: number analyzed (Participants) | 20 | 21
  Day 366 | 291.8 [149.2 to 570.4] | 301.0 [163.3 to 554.8]

25. Secondary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351 for Arms 2A and 2B
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351
Time Frame: Day 1 Pre-Dose, Day 29, Day 57, Day 85, Day 147, Day 237, Day 422
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351
Number analyzed (Participants) | 5 | 6
Titer
  Day 1, Pre-Dose | 12.1 [4.1 to 35.7] | 5.8 [4.0 to 8.4]
  Day 29 | 129.9 [5.5 to 3085.5] | 18.0 [2.5 to 130.1]
  Day 57 | 518.4 [147.9 to 1817.0] | 163.9 [58.9 to 456.1]
  Day 85 | 670.9 [321.2 to 1401.5] | 298.6 [135.7 to 657.1]
  Day 147 | 298.3 [144.1 to 617.7] | 105.5 [63.2 to 176.0]
  Day 237 | 106.3 [32.2 to 351.0] | 30.6 [24.6 to 38.1]
  Day 422: number analyzed (Participants) | 5 | 5
  Day 422 | 275.5 [28.6 to 2650.4] | 382.2 [51.3 to 2847.2]

26. Secondary Outcome: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351 for Arms 2C-H
Description: Geometric Mean (GM) of Pseudovirus Neutralization Against B.1.351. Arms 2C and 2G Day 43 samples were used for pseudovirus neutralization assay validation and results included for completeness. Samples for other vaccination groups at Day 43 were not tested for neutralization.
Time Frame: Day 1 Pre-Dose, Day 29, Day 43, Day 57, Day 119, Day 209, Day 394
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 12 | 13 | 13 | 12 | 13 | 12
Titer
  Day 1, Pre-Dose | 10.1 [3.4 to 30.3] | 6.3 [4.7 to 8.4] | 7.7 [5.4 to 10.9] | 7.4 [5.0 to 10.9] | 7.0 [5.1 to 9.7] | 14.5 [3.8 to 55.1]
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 11 | 12 | 12
  Day 29 | 40.7 [12.7 to 130.2] | 25.4 [10.2 to 63.2] | 51.9 [12.5 to 215.2] | 44.9 [10.1 to 200.1] | 51.6 [19.1 to 139.0] | 132.5 [31.0 to 567.6]
  Day 43: number analyzed (Participants) | 10 | 0 | 0 | 0 | 0 | 0
  Day 43 | 1711.4 [1031.9 to 2838.2] |  |  |  |  |
  Day 57: number analyzed (Participants) | 12 | 12 | 12 | 10 | 12 | 12
  Day 57 | 918.5 [612.6 to 1377.3] | 916.8 [654.0 to 1285.3] | 589.8 [284.7 to 1222.0] | 338.3 [145.5 to 786.5] | 946.7 [541.2 to 1656.2] | 1435.4 [651.7 to 3161.3]
  Day 119: number analyzed (Participants) | 12 | 12 | 11 | 10 | 9 | 12
  Day 119 | 386.2 [277.7 to 537.1] | 404.5 [277.7 to 589.1] | 348.9 [168.7 to 721.9] | 214.7 [83.5 to 551.8] | 479.0 [188.3 to 1218.1] | 643.1 [274.5 to 1506.7]
  Day 209: number analyzed (Participants) | 11 | 12 | 12 | 9 | 9 | 11
  Day 209 | 164.0 [84.2 to 319.6] | 138.4 [84.4 to 226.9] | 137.9 [65.3 to 291.5] | 75.4 [30.4 to 186.9] | 133.1 [55.0 to 322.0] | 170.6 [50.5 to 576.2]
  Day 394: number analyzed (Participants) | 11 | 9 | 8 | 10 | 8 | 9
  Day 394 | 1281.6 [449.8 to 3651.4] | 341.1 [72.2 to 1611.8] | 1006.9 [359.8 to 2818.0] | 671.1 [286.9 to 1569.9] | 1609.1 [276.9 to 9349.4] | 2349.3 [1024.0 to 5389.8]

27. Secondary Outcome: Number of Participants Who Seroconverted Against D614G for Arms 1A and 1B
Description: Number of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from baseline against D614G.
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 366
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23
Participants
  Day 15 | 24 | 23
  Day 29 | 24 | 23
  Day 91 | 25 | 23
  Day 181: number analyzed (Participants) | 22 | 23
  Day 181 | 19 | 21
  Day 366: number analyzed (Participants) | 20 | 22
  Day 366 | 12 | 12

28. Secondary Outcome: Number of Participants Who Seroconverted Against D614G for Arms 2A and 2B
Description: as for outcome 27
Time Frame: Day 29, Day 57, Day 85, Day 147, Day 237, Day 422
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351
Number analyzed (Participants) | 5 | 6
Participants
  Day 29 | 5 | 4
  Day 57 | 5 | 6
  Day 85 | 5 | 6
  Day 147 | 5 | 6
  Day 237 | 4 | 5
  Day 422: number analyzed (Participants) | 5 | 5
  Day 422 | 3 | 5

29. Secondary Outcome: Number of Participants Who Seroconverted Against D614G for Arms 2C-H
Description: Number of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from baseline against D614G. Arms 2C and 2G Day 43 samples were used for pseudovirus neutralization assay validation and results included for completeness. Samples for other vaccination groups at Day 43 were not tested for neutralization.
Time Frame: Day 29, Day 43, Day 57, Day 119, Day 209, Day 394
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 12 | 13 | 13 | 12 | 13 | 12
Participants
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 11 | 12 | 12
  Day 29 | 3 | 3 | 12 | 11 | 11 | 7
  Day 43: number analyzed (Participants) | 10 | 0 | 0 | 0 | 12 | 0
  Day 43 | 10 |  |  |  | 12 |
  Day 57: number analyzed (Participants) | 12 | 12 | 12 | 10 | 12 | 12
  Day 57 | 11 | 12 | 12 | 10 | 12 | 12
  Day 119: number analyzed (Participants) | 12 | 12 | 11 | 10 | 9 | 12
  Day 119 | 11 | 12 | 11 | 10 | 9 | 12
  Day 209: number analyzed (Participants) | 11 | 12 | 12 | 9 | 9 | 11
  Day 209 | 10 | 11 | 11 | 9 | 8 | 10
  Day 394: number analyzed (Participants) | 11 | 9 | 8 | 10 | 8 | 9
  Day 394 | 11 | 8 | 7 | 10 | 8 | 8

30. Secondary Outcome: Number of Participants Who Seroconverted Against B.1.351 for Arms 1A and 1B
Description: Number of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from baseline against B.1.351.
Time Frame: Day 15, Day 29, Day 91, Day 181, Day 366
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: 50 mcg of mRNA-1273.351 | 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 25 | 23
Participants
  Day 15 | 25 | 23
  Day 29 | 25 | 23
  Day 91 | 25 | 23
  Day 181: number analyzed (Participants) | 22 | 23
  Day 181 | 22 | 20
  Day 366: number analyzed (Participants) | 20 | 21
  Day 366 | 18 | 15

31. Secondary Outcome: Number of Participants Who Seroconverted Against B.1.351 for Arms 2A and 2B
Description: as for outcome 30
Time Frame: Day 29, Day 57, Day 85, Day 147, Day 237, Day 422
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351
Number analyzed (Participants) | 5 | 6
Participants
  Day 29 | 4 | 2
  Day 57 | 5 | 5
  Day 85 | 5 | 6
  Day 147 | 5 | 6
  Day 237 | 4 | 5
  Day 422: number analyzed (Participants) | 5 | 5
  Day 422 | 4 | 5

32. Secondary Outcome: Number of Participants Who Seroconverted Against B.1.351 for Arms 2C-H
Description: Number of participants who seroconverted defined as a 4-fold change in pseudovirus neutralization from baseline against B.1.351. Arms 2C and 2G Day 43 samples were used for pseudovirus neutralization assay validation and results included for completeness. Samples for other vaccination groups at Day 43 were not tested for neutralization.
Time Frame: Day 29, Day 43, Day 57, Day 119, Day 209, Day 394
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
Number analyzed (Participants) | 12 | 13 | 13 | 12 | 13 | 12
Participants
  Day 29: number analyzed (Participants) | 12 | 13 | 13 | 11 | 12 | 12
  Day 29 | 4 | 5 | 5 | 6 | 6 | 8
  Day 43: number analyzed (Participants) | 10 | 0 | 0 | 0 | 0 | 0
  Day 43 | 10 |  |  |  |  |
  Day 57: number analyzed (Participants) | 12 | 12 | 12 | 10 | 12 | 12
  Day 57 | 11 | 12 | 12 | 9 | 12 | 11
  Day 119: number analyzed (Participants) | 12 | 12 | 11 | 10 | 9 | 12
  Day 119 | 11 | 12 | 11 | 9 | 9 | 11
  Day 209: number analyzed (Participants) | 11 | 12 | 12 | 9 | 9 | 11
  Day 209 | 11 | 12 | 11 | 7 | 8 | 9
  Day 394: number analyzed (Participants) | 11 | 9 | 8 | 10 | 8 | 9
  Day 394 | 11 | 8 | 8 | 10 | 8 | 8

ADVERSE EVENTS:
Time Frame: Solicited (local and systemic) AEs were collected from Day 1 through Day 7 for Arms 1A-2H, Day 29 through Day 36 for Arms 2A-2H, and Day 57-64 for Arms 2A-2B. Unsolicited AEs were collected from Day 1 through Day 29 from Arms 1A-2H, Day 29 through Day 57 for Arms 2A-2H, and Day 57 through Day 85 for Arms 2A-2B. SAEs, MAAEs, and NOCMCs were collected from Day 1 through Day 366 for Arms 1A and 1B, Day 1 to Day 422 for Arms 2A and 2B, and Day 1 to Day 394 for Arms 2C-2H.
Description: Systemic AEs include headache, fatigue, myalgia, arthralgia, nausea, fever, and chills. Local events include injection site pain, injection site erythema, injection site edema/induration. Unsolicited AEs were all AEs spontaneously reported by the subject and/or in response to an open question from study staff or revealed by observation, physical examination or other diagnostic procedures.
Arm/Group | Arm 1A: 50 mcg of mRNA-1273.351 | Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 0/5 | 0/6 | 0/12 | 0/13 | 0/13 | 0/12 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/23 | 0/5 | 0/6 | 0/12 | 0/13 | 0/13 | 0/12 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 24/25 | 23/23 | 5/5 | 6/6 | 12/12 | 12/13 | 13/13 | 11/12 | 13/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1A: 50 mcg of mRNA-1273.351 (N=25) | Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 (N=23) | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 (N=5) | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 (N=6) | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 (N=12) | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 (N=13) | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 (N=13) | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 (N=12) | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 (N=13) | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 (N=13)
Paresthesia of upper extremity (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1A: 50 mcg of mRNA-1273.351 (N=25) | Arm 1B: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 (N=23) | Arm 2A: 100 mcg mRNA-1273/100 mcg mRNA-1273/50 mcg mRNA-1273.351 (N=5) | Arm 2B: 50 mcg mRNA-1273/50 mcg mRNA-1273/50 mcg mRNA-1273.351 (N=6) | Arm 2C: 100 mcg mRNA-1273.351/100 mcg mRNA-1273.351 (N=12) | Arm 2D: 50 mcg mRNA-1273.351/50 mcg mRNA-1273.351 (N=13) | Arm 2E: 100 mcg mRNA-1273/100 mcg mRNA-1273.351 (N=13) | Arm 2F: 50 mcg mRNA-1273/50 mcg mRNA-1273.351 (N=12) | Arm 2G: 50 mcg mRNA-1273 + 50 mcg mRNA-1273.351/50 mcg mRNA-1273 + 50 mcg mRNA-1273.351 (N=13) | Arm 2H: 25 mcg mRNA-1273 + 25 mcg mRNA-1273.351/25 mcg mRNA-1273 + 25 mcg mRNA-1273.351 (N=13)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Athletic heart syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraclavicular fossa pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 1 (1) | 0
Swelling (General disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (2)
COVID-19 (Infections and infestations) | 2 (2) | 4 (4) | 0 | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1)
Blood cholesterol increased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1)
Burning sensation (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 0
Headache (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Depression (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 6 (6) | 9 (9) | 2 (3) | 1 (1) | 6 (6) | 2 (3) | 5 (6) | 3 (3) | 5 (7) | 4 (5)
Chills (General disorders) | 17 (17) | 10 (10) | 4 (7) | 5 (6) | 7 (9) | 4 (4) | 6 (11) | 4 (5) | 8 (9) | 6 (6)
Fatigue (General disorders) | 22 (22) | 19 (19) | 5 (11) | 5 (8) | 9 (14) | 11 (19) | 12 (20) | 9 (15) | 10 (14) | 11 (17)
Pyrexia (General disorders) | 6 (6) | 5 (5) | 3 (4) | 1 (1) | 4 (5) | 1 (1) | 3 (3) | 0 | 2 (2) | 2 (2)
Vaccination site erythema (General disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 2 (3) | 3 (4) | 2 (2) | 2 (2) | 4 (5) | 3 (3)
Vaccination site induration (General disorders) | 5 (5) | 2 (2) | 2 (5) | 0 | 2 (4) | 2 (2) | 3 (3) | 1 (1) | 6 (6) | 5 (7)
Vaccination site pain (General disorders) | 24 (24) | 20 (20) | 5 (12) | 6 (17) | 10 (18) | 12 (23) | 13 (22) | 11 (20) | 12 (22) | 13 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 6 (6) | 4 (8) | 2 (2) | 5 (5) | 7 (8) | 5 (7) | 2 (3) | 4 (6) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (17) | 20 (20) | 4 (6) | 5 (8) | 8 (9) | 10 (13) | 9 (14) | 8 (11) | 10 (14) | 8 (10)
Headache (Nervous system disorders) | 19 (19) | 12 (12) | 3 (7) | 5 (6) | 10 (12) | 9 (13) | 11 (18) | 7 (9) | 9 (15) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (4):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT04785144/Prot_001.pdf
  • Statistical Analysis Plan: 21-0002_SAP1 (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT04785144/SAP_002.pdf
  • Statistical Analysis Plan: 21-0002_SAP2 (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT04785144/SAP_003.pdf
  • Informed Consent Form (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT04785144/ICF_004.pdf